CLINICAL TRIAL: NCT03970421
Title: Demographic and Clinical Data Associated to Head Injury Severity on Adults Patients (Older Than 16yo), and Follow up for 90 Days to Check the Development of Associated Complications, Deciding the Optimal Observation Lapse at ED
Brief Title: Severity Factors and Needed Observation Time at ED of Patients Wih Head Injury
Acronym: HESCTCE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital El Escorial (Other)
Responsible Party: Sponsor
Other Study IDs: URGHESCHEADINJURY
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Head Injury Other; Length of Stay; Delayed Complications
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- patients without anticoagulant and / or antiplatelet treatment: Patients older than 16yo with no anticoagulant or antiplatelet treatment attended at ED because of Head Injury and with a Head CT performed.
  Interventions: Other: Observation
- patients on antiplatelet therapy (ASA and / or clopidogrel: Patients older than 16yo on antiplatelet treatment attended at ED because of Head Injury and with a Head CT performed.
  Interventions: Other: Observation
- patients on treatment with acenocoumarol and INR <2: Patients older than 16yo on acenocumarol and with INR <2 attended at ED because of Head Injury and with a Head CT performed.
  Interventions: Other: Observation
- Others: patients on anticoagulant therapy with acenocoumarol and INR> = 2 or patients on treatment with direct thrombin inhibitors (dabigatran), or inhibitors of factor Xa (rivaroxaban, apixaban, edoxaban) or patients on treatment with low molecular weight heparins (LMWH) attended at ED because of Head Injury and with a Head CT performed.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Check clinical status at different time intervals during 3 months

SUMMARY:
We know precisely which patients and when they should have an imaging test to evaluate a Head Injury (HI). But in those patients on anticoagulant and / or antiaggregant treatment we do not know the exact incidence of early and late hemorrhagic lesions, and there is no specific recommendation on how long they should remain under observation in the emergency department if no initial lesions are evident. Our goal is to try to answer these two questions.

DETAILED DESCRIPTION:
MATERIAL: Prospective study of patients treated of HI in the Emergency Department (ED) and to whom an image test is performed (cranial CT scan). Collection of demographic, clinical, analytical, image tests, and observation time in the emergency department (from admission to medical discharge)

METHODS: Separation of subjects included in the study in 4 cohorts: patients without anticoagulant and / or antiaggregant treatment; patients with antiplatelet therapy (ASA and / or clopidogrel); patients with anticoagulant treatment with acenocoumarol and INR <2; and patients on anticoagulant therapy with acenocoumarol and INR> = 2 or patients on treatment with direct thrombin inhibitors (dabigatran), or inhibitors of factor Xa (rivaroxaban, apixaban, edoxaban) or patients on treatment with low molecular weight heparins (LMWH) ) Follow-up through analysis of clinical history and telephone interview at 2, 7, 15, 30, 60 and 90 days.

Statistical analysis of the results.

ELIGIBILITY:
Inclusion Criteria:

* HI attended at ED
* Head CT performed as recommended by clinical guides
* Contact data available (phone number)

Exclusion Criteria:

* Patients not able for follow up (foreigners or tourists or whatsoever whom are not going to stay on the country for at least 3 months)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated by HI in the Emergency Department (ED) and to whom an imaging test is performed (cranial CT scan)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Severity factors associated to head injury | 24 hours
  Demographical, clinical, analitical, and neuroimaging data associated to severity of HI
Development of haemorragical complications during observation time | 90 days
  Finding of an haemorragical injury associated with the head injury during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Favá, PhD, Study Chair — Hospital El Escorial
Locations (1):
- Hospital EL Escorial, El Escorial, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No